CLINICAL TRIAL: NCT02887131
Title: Evaluation of Dynamic Computed Tomography Anatomy of Ankle in Inversion / Eversion Mouvement in Subtalar Instability.
Brief Title: Dynamic Imaging of the Subtalar Instability
Acronym: IDIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PSS 2011/IDIS-LUX/NK
Record Dates: First submitted 2012-02-29; First posted 2016-09-02 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Subtalar Arthritis; Subtalar Instability
Keywords: Subtalar arthritis; Subtalar instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy volunteers (Experimental)
  Interventions: Other: Dynamic CT of the ankle
- Arthritis (Experimental)
  Interventions: Other: Dynamic CT of the ankle
- Instability (Experimental)
  Interventions: Other: Dynamic CT of the ankle

INTERVENTIONS:
Other: Dynamic CT of the ankle — during inversion and eversion mouvement, with Aquilion One Toshiba scanner

SUMMARY:
The purpose of this study is to describe normal dynamic computed tomography anatomy of hind foot in inversion/eversion movement, and to define diagnostic criteria for subtalar instability.

DETAILED DESCRIPTION:
Dynamic CT (Aquilion One Toshiba) of the ankle during inversion and eversion movement will be performed in patients from three groups: healthy volunteers, patients with subtalar arthritis, and patients with suspicion of subtalar instability.

ELIGIBILITY:
Inclusion Criteria:

* Group Instability: suspicion of subtalar instability
* Group Arhtritis: subtalar stiffness
* Group Healthy volunteers: healthy volunteers
* conscious and cooperating
* written consent obtained after oral and written clear and intelligible information
* no pregnancy

Exclusion Criteria:

* pregnancy
* unable to understand information about this study
* unable to understand the movement of inversion / eversion of ankle
* absence of affiliation to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Talocalcaneal angle | baseline
Maximum exposed distance on superolateral surface of calcaneum | baseline
Minimum distance between sustentaculum tali and talus posteromedial tubercle | baseline
Maximum distance between sustentaculum tali and talus posteromedial tubercle | baseline
Maximum anterolateral talocalcaneal distance | baseline
Maximum posterolateral talocalcaneal distance | baseline
Minimum posterolateral talocalcaneal distance | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital, Nancy, France, France

IPD SHARING:
Plan to Share IPD: No